CLINICAL TRIAL: NCT06536985
Title: Effect of an Oral Frailty Measures Program in Institutionalized Elders: a Study Protocol of a Cluster-Randomized Controlled Trial
Brief Title: Effect of an Oral Frailty Measures Intervention Programs in Institutionalized Elders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, HangTian Zhu, Principal Investigator, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024100
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Frailty
Keywords: Nursing Homes; Aged; Exercise
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The first author will use randomizer.org for randomization. Recruitment without informing the subjects of study participation and group allocation to blind the subjects. And the allocation is also concealed for researchers in charge of data collection and processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contral group (Active Comparator)
  Interventions: Behavioral: Contral group
- Treatment group (Experimental)
  Interventions: Behavioral: treatment group

INTERVENTIONS:
Behavioral: treatment group — Researchers will collaborate with participants to develop personalized intervention plans, which include physical exercise, oral function training, basic dietary guidance, and detailed oral health knowledge directly related to oral health behaviors. To facilitate better communication and management, a WeChat group will be created to encourage participants to share their daily exercise achievements. In the first week, face-to-face oral function training sessions will be organized for the intervention group at the nursing home activity center. Concurrently, once a week, the intervention group will gather at the nursing home activity center to practice together using illustrated videos. On Wednesdays, educational articles and videos about oral health are sent via text message. On Fridays, a group communication activity is organized to enhance their social connections. Additionally, we will guide elderly participants to master essential internet skills, enabling them to use smartphones to
  Arms: Treatment group
Behavioral: Contral group — Participants in the control group will receive general lifestyle advice via text message once or twice a week.They will not participate in the intervention's fitness routines, online classes, group chats, or films with health educators. Individual workout regimens, goals, or comments are not given by researchers. Participants in the control group's complaints or questions will always be answered with basic health information and suggestions. Researchers won't ask for individual advice or comments from other professionals.
  Arms: Contral group

SUMMARY:
This is a compelling 16-week prospective, double-blind, whole-cluster randomized controlled trial(RCT).This study will recruit 226 older adults over the age of 65.Based on King's goal attainment theory, a program to promote oral health is developed.The study aims to evaluate the effectiveness of a mixed face-to-face and eHealth oral health promotion program for older adults with oral frailty in nursing homes, based on the Theory of Planned Behavior.

DETAILED DESCRIPTION:
Background:

Oral frailty is a progressive loss of oral function associated with aging, usually caused by a variety of injuries. Some recent studies have shown that oral frailty is closely linked to physical functioning (physical frailty and changes in body composition), as well as nutritional status (low protein intake, poor dietary diversity, and malnutrition) in older adults in addition, a significant association between inadequate social network participation and poor oral function has also been confirmed by research. Oral frailty in older adults not only decreases their quality of life but also leads to serious problems like cognitive impairment, falls, disability, and even death. This puts a strain on families and society in terms of healthcare. Early Identifying and treating oral frailty is important for improving the quality of life of older adults and reducing the pressure on healthcare resources.

Aim:

The researchers hypothesize that a health program based on King's goal achievement theory will have a significant effect on oral frailty among older adults in nursing homes. Therefore, in this study, researchers will explore the impact of a health program based on King's goal achievement theory on oral frailty in older adults residing in nursing homes.

Methods:

This is a compelling 16-week prospective, double-blind, whole-cluster randomized controlled trial designed to evaluate a program aimed at enhancing oral health in older adults residing in nursing homes who experience oral frailty. The program combines in-person and online activities, aligning with the goal attainment theory. Once a week, the intervention group gathers at the nursing home activity center to practice together using illustrated videos. On Wednesdays, educational articles and videos about oral health are sent via text message. On Fridays, a group communication activity is organized to enhance their social connections. Additionally, we will guide the elderly participants to master essential internet skills, use smartphones to stay in touch with friends and family, and provide timely feedback on issues through smartphones. Any reports or inquiries received through any channel will be promptly addressed.

Participants and demographic data:

Researchers will recruit patients with oral frailty from two welfare institutions in Hangzhou City in the following three main ways:1. Public information sessions: Information sessions were held in the activity centers of the nursing facilities to introduce the study to potential participants and encourage their participation.

2. Local advertising: Posters and flyers were placed in the nursing facilities.3. Online recruitment: Recruitment information was posted using social media (WeChat), professional forums, and other online channels.

Procedure and Data collection:

This is a compelling 16-week prospective, double-blind, whole-cluster randomized controlled trial. The study adheres to the ethical principles of the Helsinki Declaration and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) checklist. It has been approved by the Medical Ethical Committee of Hangzhou Normal University（Ratification date is September 14 2024, 2024100）

Statistical analysis:

We used repeated measures two-way ANOVA to determine the effectiveness of independent intervention variables. The independent variables were group (intervention/control) and time (baseline/week 12). The dependent variable was the oral frailty measure. We examined the effects of program continuation using repeated measures two-way ANOVA and conducted post hoc testing using Bonferroni methods. All statistical analyses were performed using IBM SPSS Statistics for Windows version 24.0 (IBM Corp., Armonk, NY, USA). Statistically significant differences were defined as p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old
2. Residing in a nursing home for ≥ 3 months
3. Meeting at least three of the six criteria for oral frailty
4. Conscious and with normal reading and comprehension abilities
5. Informed consent to participate in this study

Exclusion Criteria:

1. Edentulous state without dentures
2. Cognitive or communication impairments
3. Elderly lacking self-care ability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Assessing changes in the risk of oral frailty | Before and 16 weeks after the intervention
  Oral frailty risk was assessed using the Chinese version of the Oral Frailty Index-8 (OFI-8 scale) translated by zongme.The scale consists of eight items with a total score ranging from 0 to 11, with higher scores indicating poorer oral health and higher risk of oral frailty. These include healthy (0-2 points), pre oral debilitation (3 points), oral debilitation (4-6 points) and severe oral debilitation (≥7 points).
Assessing changes in oral function status | Before and 16 weeks after the intervention
  We will use the Oral Frailty Assessment Instrument (OFI) created by Tanaka to measure the presence or absence of oral frailty and the detailed status of oral functioning to provide a basis for targeted interventions at a later stage. An assessment was made based on 6 items in the method described by Tanaka et al. These included the number of teeth, mastectomy function, articulation skills, tongue pressure, subjective feeding, and swallowing difficulty or not. Oral fragility was considered exist if at least 3 of the criteria were met. These included (1) Lower number of remaining teeth;(2) mastectomy score; (3) oral motor skills; (4) tongue pressure; (5) eating hard foods with subjective difficulty (yes); and (6) subjective dysphagia (yes). We used the Kihon questionnaire to ask about any difficulties with eating hard food and swallowing.

SECONDARY OUTCOMES:
Assessment of changes in body composition | Before and 16 weeks after the intervention
  Participants will have body composition measured by using bioelectrical impedance analysis (BIA) with InBody 720 device.Detection content including: body weight (kg), skeletal muscle mass (kg), body fat mass (kg), BMI (kg/m2), body fat percentage (%) and waist--to--hip ratio).Participants will be told not to exercise for at least 24 hours before the test, not to consume alcohol or excessive amounts of caffeine, and not to eat and drink for four hours before the test, but water can be consumed up to 45 minutes before the test.
Nutrition Screening | Before and 16 weeks after the intervention
  We will use the Mini-Nutritional Assessment Short Form (MNA-SF) to assess the nutritional status of older adults in nursing facilities. The scale was created by Rubenstein et al. and includes six assessment categories: changes in food intake over the past three months, changes in body weight, mobility, acute illness or injury, psychosomatic problems, and body mass index (BMI). The scale goes up to 14 points. A score of 11 or higher is normal, while a score below 11 might indicate a risk of malnutrition. The Cronbach's alpha coefficient was 0.833, showing that the scale is reliable for assessing the nutritional status of elderly people because it has a high internal consistency.
Changes in Social Support | Before and 16 weeks after the intervention
  We will use the The Multidimensional Scale of Perceived Social Suppor（MSPSS） to measure social support levels. It was developed by Ziniet and revised by Keeley Zhou in China. There are three dimensions, including family support, other people's support, and friends' support. The scale was scored on a 7-points Likert scale, with a total score of 12-84 points. According to the total scores of the scale, comprehension of social support was categorized into 3 levels, with 12-36 points as low level, 37-60 points as medium level, and 61-84 points as high level.
Self Efficacy | Before and 16 weeks after the intervention
  In this study, the Geriatric Self⁃Efficacy Scale for Oral Health (GSEOH) will be used to identify the current status of oral health self-efficacy of the subjects, which was developed by Ohara, et al. The GSEOH has 3 dimensions and 20 items. These dimensions are oral function (9 items) and oral health. They were developed by the University of California, Los Angeles. The scale has three dimensions and a total of 20 items. These dimensions are oral function (9 items), oral hygiene habits (8 items), and oral consultation habits (3 items). The scale uses a 4-point Likert scale, with 1 meaning "not confident" and 4 meaning "very confident". The total scores can range from 20 to 80 points, or from 1 to 4 points. The higher the scores, the higher the oral health-related self-efficacy of the elderly.
Changes in frailty | Before and 16 weeks after the intervention
  The Groningen Frailty Indicator Scale will be used in this study to determine if patients are frail or not. The scale was developed by the Dutch scholar Steverink , and translated by Xiang Wei Frailty Scale, which evaluates the patients from multiple dimensions, including 4 dimensions of somatic, cognitive, psychological and social. Each of these entries is scored as "0" or "1" according to the score, and the total score ranges from 0 to 15. A larger score indicates a more severe degree of debilitation in the patient. The original scale uses a threshold value of 4. Patients with a score above 4 are considered debilitated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No